CLINICAL TRIAL: NCT01362725
Title: Spinal Cord Stimulation For Heart Failure As A Restorative Treatment
Brief Title: Spinal Cord Stimulation For Heart Failure
Acronym: SCS HEART
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-10-029-ID-SC
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Systolic Heart Failure
Keywords: spinal cord stimulation; systolic heart failure
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal cord stimulation (Experimental)
  Interventions: Device: Spinal cord stimulation system

INTERVENTIONS:
Device: Spinal cord stimulation system — An implantable pulse generator (IPG) will deliver low-intensity electrical pulses which travel from the IPG through the leads to the electrodes positioned at the selected nerve fibers to provide the therapeutic stimulation.
  Other Names: Eon Mini Neurostimulation System,; Octrode® percutaneous lead (Model 3186),; Eon Mini IPG (Model 3788),; Eon Patient ProgrammerTM (Model 3851),; Multi-program trial stimulator (Model 3510),; Rapid programmer (Model 3832),; Eon Mini Charging System (Model 3721).; Similar St. Jude Medical commercially available neurostimulation system with the same capabilities may also be used.

SUMMARY:
The primary objectives of this feasibility study are to determine the safety of spinal cord stimulation (SCS) as a therapy in patients with systolic heart failure and to gather observational information for potential efficacy markers

DETAILED DESCRIPTION:
Morbidity and mortality in heart failure patients remain relatively high, even with recent advances in therapies. Previous studies show that the autonomic nervous system plays an important role in the pathophysiology of heart failure (HF)and sudden cardiac death.

SCS is a neurostimulation therapy, which involves the stimulation of selected nerve fibers and intends to create end-organ responses characterized by changes in blood flow, decrease of catecholamines and reduction in inflammation. These changes that occur due to SCS are shown to be effective in reducing the symptoms of chronic angina and pain secondary to peripheral vascular disease where both situations are characterized by decreased blood flow and inflammation.

The SCS system consists of an implantable pulse generator(IPG) and lead(s). Each lead has electrodes on the distal end. Electrical impulses travel from the IPG through the leads to the electrodes positioned at the selected nerve fibers to provide the therapeutic stimulation. By virtue of its potential in augmenting blood flow, decreasing catecholamines and reducing inflammation, SCS may further benefit patients with heart failure (HF).

ELIGIBILITY:
Inclusion Criteria:

* Patients has a LVEF between 20% and 35%
* Patient is in NYHA Class III or in Ambulatory Class IV
* Patient has had a SJM implantable cardioverter defibrillator (ICD) device or a SJM CRT-D device implanted >90 days and is receiving stable medical therapy for HF (>90 days) at Baseline
* Patient has a LV end diastolic diameter between 55mm and 80mm
* Patient must be able and willing to provide written informed consent to participate in this study
* Patient must be able and willing to comply with the required follow-up schedule

Exclusion Criteria:

* Patient currently has an implanted spinal cord stimulator or previously had an implanted spinal cord stimulator which is now explanted
* Patient has polyneuropathy
* Patient requires short-wave diathermy, microwave diathermy or therapeutic ultrasound diathermy
* Patient has received a tissue / organ transplant (or is expected to have a tissue / organ transplant within the next 180 days)
* Patient has persistent or permanent Atrial Fibrillation (AF)
* Patient has chronic refractory angina or peripheral vascular pain
* Patient has critical valvular heart disease that requires valve repair or replacement
* Patient has had a myocardial infarction (MI) or cardiac revascularization procedure(percutaneous coronary intervention or coronary artery bypass graft) <90 days at Baseline or is expected to have this in the next 180 days
* Patient is on IV inotropic therapy
* Patient has active myocarditis or early postpartum cardiomyopathy
* Patient has taken any of the following drugs within 30 days of enrollment: systemic corticosteroids, cytostatic and immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), DNA depleting or cytotoxic drugs
* Patient is pregnant, or of childbearing potential and is not using adequate contraceptive methods, or nursing
* Patient with a bleeding tendency (International Normalized Ratio, INR >1.2 and platelet count <100 x109 per liter)
* Patient has a local infection at the ICD implant location or systemic infection
* Patient has renal insufficiency (creatinine >3.0 mg/dl)
* Patient is participating in another clinical study
* Patient is less than 18 years old
* Patient's life's expectancy is less than 1 year as assessed by investigators

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2014-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy markers | 6 months
  Intra and post procedure adverse events, exercise and functional capacity, left ventricular structure and function, inflammatory condition, and quality of life.

SECONDARY OUTCOMES:
long-term safety | 24 months
  post procedural adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Fat Tse, MD, Principal Investigator — The University of Hong Kong, Queen Mary Hospital
Locations (5):
- Australia (2):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan (2):
  - Osaka University Hospital, Osaka
  - University of Tokyo Hospital, Tokyo

REFERENCES:
- [Background] Lopshire JC, Zhou X, Dusa C, Ueyama T, Rosenberger J, Courtney N, Ujhelyi M, Mullen T, Das M, Zipes DP. Spinal cord stimulation improves ventricular function and reduces ventricular arrhythmias in a canine postinfarction heart failure model. Circulation. 2009 Jul 28;120(4):286-94. doi: 10.1161/CIRCULATIONAHA.108.812412. Epub 2009 Jul 13. PMID 19597055
- [Background] Foreman RD, Linderoth B, Ardell JL, Barron KW, Chandler MJ, Hull SS Jr, TerHorst GJ, DeJongste MJ, Armour JA. Modulation of intrinsic cardiac neurons by spinal cord stimulation: implications for its therapeutic use in angina pectoris. Cardiovasc Res. 2000 Aug;47(2):367-75. doi: 10.1016/s0008-6363(00)00095-x. PMID 10946073
- [Background] Armour JA, Linderoth B, Arora RC, DeJongste MJ, Ardell JL, Kingma JG Jr, Hill M, Foreman RD. Long-term modulation of the intrinsic cardiac nervous system by spinal cord neurons in normal and ischaemic hearts. Auton Neurosci. 2002 Jan 10;95(1-2):71-9. doi: 10.1016/s1566-0702(01)00377-0. PMID 11873770
- [Background] Deer TR, Raso LJ. Spinal cord stimulation for refractory angina pectoris and peripheral vascular disease. Pain Physician. 2006 Oct;9(4):347-52. PMID 17066119
- [Background] Mannheimer C, Carlsson CA, Emanuelsson H, Vedin A, Waagstein F, Wilhelmsson C. The effects of transcutaneous electrical nerve stimulation in patients with severe angina pectoris. Circulation. 1985 Feb;71(2):308-16. doi: 10.1161/01.cir.71.2.308. PMID 3871177
- [Derived] Tse HF, Turner S, Sanders P, Okuyama Y, Fujiu K, Cheung CW, Russo M, Green MDS, Yiu KH, Chen P, Shuto C, Lau EOY, Siu CW. Thoracic Spinal Cord Stimulation for Heart Failure as a Restorative Treatment (SCS HEART study): first-in-man experience. Heart Rhythm. 2015 Mar;12(3):588-595. doi: 10.1016/j.hrthm.2014.12.014. Epub 2014 Dec 12. PMID 25500165